CLINICAL TRIAL: NCT03900936
Title: Detecting Dementia Earlier: Using Spatial & Episodic Memory Tests to More Accurately Predict Progression From Mild Cognitive Impairment to Alzheimer's Disease
Brief Title: Detecting Dementia Earlier
Acronym: DDE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: South Tees Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 207985
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Alzheimer Disease; MCI; Aging
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neuropsychological tests: This study is not an intervention as such. We are simply comparing the scores of MCI patients who subsequently went on to develop dementia vs those who did not.
  Interventions: Diagnostic Test: Neuropsychological tests

INTERVENTIONS:
Diagnostic Test: Neuropsychological tests — This study is not an intervention as such. We are simply comparing the scores of MCI patients who subsequently went on to develop dementia vs those who did not.

SUMMARY:
Aims

1. To determine whether the 4 Mountains test of allocentric (i.e. viewpoint-independent) spatial memory, and tests of memory for a recent experience (e.g. watching a brief video), to diagnose the early stages of Alzheimer's disease.
2. We operationalise this as the ability of these tests to predict whether or not an individual progresses from having some cognitive difficulties (diagnosed as 'mild cognitive impairment' MCI) to subsequently developing Alzheimer's disease up to two years later.
3. To assess whether the ability to diagnose early stages of Alzheimer's disease can be improved by combining the scores from different memory tests, from questionnaires assessing spatial and social aspects of everyday life.
4. To assess whether scores on the spatial memory test are correlated with patients' reports of their everyday spatial memory, using a newly-developed questionnaire.

Outcome Measures

Primary study objective:

To determine the ability of allocentric spatial and episodic memory test performance to predict progression from mild cognitive impairment (MCI) to Alzheimer's disease.

Secondary outcome measure

1. To assess to what extent social characteristics of everyday life may impact upon progression from mild cognitive impairment (MCI) to Alzheimer's disease.
2. To correlate allocentric spatial test performance with real-world spatial ability as assessed through a novel spatial questionnaire.

DETAILED DESCRIPTION:
In recent years, the need for tests that reliably diagnose the early stages of Alzheimer's disease (AD) with high accuracy has been strongly emphasised. Detecting AD in its earliest stages increases the likelihood that therapeutic agents (e.g. newly-developed drugs) and interventions (e.g. changes in diet and exercise) can prolong the period of high-quality, independent living and reduce the impact on patients, families and care providers. An ideal test would have the sensitivity to detect everyone who has early-stage AD, while simultaneously not giving a 'false alarm' to anyone who shows some age-related impairments in cognition but who does not have early-stage AD. Secondly, an ideal test should be free and simple to administer on a national scale, without requiring extensive training on the part of the testers to set up, run, and interpret. Unfortunately, currently used tests do not come close to this ideal. There are some good biomarker-based tests for early stages of AD, but they are costly, highly invasive and in effect impossible to use for national screening purposes. MRI imaging of brain regions affected early in AD detects early AD no better than neuropsychological testing and whilst it is non-invasive, many patients find it aversive. Here, we propose to examine whether the use of spatial and episodic memory tests can get us nearer to this ideal, whether used singly, together, or in combination with other tests.

The project has two stages. In stage 1, we will administer recently-developed spatial and episodic memory tests (along with more established neuropsychological tests) to patients who have recently been diagnosed with Mild Cognitive Impairment (MCI). At stage 2, clinical follow up (c.15-30 months after MCI diagnosis) we will establish those patients who have, and have not, progressed to AD. Analysis will then determine which tests at stage 1 best predicted progression-to-AD at stage 2.

ELIGIBILITY:
Inclusion Criteria:

* . MCI diagnosis.

Exclusion Criteria:

* 1. Presence of significant neurological condition such as Traumatic Brain Injury, Epilepsy, Stroke, Multiple Sclerosis, Brain tumour, Encephalitis, Meningitis, Parkinson's disease or visual impairment severe enough to hamper processing of visual test stimuli.

  2. Major psychiatric disorder, such as schizophrenia, bipolar disorder and personality disorders such as borderline personality disorder. We will exclude severe (but not mild or moderate) clinical depression, and will exclude severe (but not mild or moderate) anxiety.

  3. The use of cognitive enhancing drugs e.g. Cholinesterase inhibitors. 4. A history of alcohol excess or excess of illicit drug use within the last 5 years.

(By definition, the diagnosis of dementia excludes a participant, since this would conflict with the fourth basis for the MCI diagnosis)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with mild cognitive impairment (MCI) will be recruited from memory clinics from several different trusts, including NHS South Tees NHS FT and NHS Tees, Esk and Wear Valleys NHS FT.
  The diagnosis of MCI will be made by clinicians in accordance with the four core clinical criteria of Albert et al (2011). Briefly, these are: 1) Evidence of change (worsening) in cognition; 2) Impairment in one or more cognitive domains greater than expected for age/education; 3) Preservation of independence in functional abilities; 4) No current dementia.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-01-19 (Actual); Primary Completion 2019-06-20 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Predicting progression | 3 years
  To determine the ability of allocentric spatial and episodic memory test performance to predict progression from mild cognitive impairment (MCI) to Alzheimer's disease.
Social Characteristics and questionnaires | 3 years
  1. To assess to what extent social characteristics of everyday life may impact upon progression from mild cognitive impairment (MCI) to Alzheimer's disease.
  2. To correlate allocentric spatial test performance with real-world spatial ability as assessed through a novel spatial questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- South Tees Hospitals NHS FT, Middlesbrough, Teesside, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
To be discussed with research team